CLINICAL TRIAL: NCT00055536
Title: A Phase II, Multi-Center, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, and Efficacy of Intravenous Antegren (Natalizumab) in Crohn's Disease Subjects Concurrently Receiving Remicade (Infliximab) and Not in Remission
Brief Title: Safety and Efficacy of Natalizumab in Combination With Remicade in the Treatment of Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD306
Record Dates: First submitted 2003-03-04; First posted 2003-03-06 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Natalizumab

INTERVENTIONS:
Drug: natalizumab

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of natalizumab in individuals diagnosed with active Crohn's Disease that are not in remission (CDAI greater than/equal to 150) and are currently taking Remicade. It is thought that natalizumab may stop the movement of certain cells, known as white blood cells, into bowel tissue. These cells are thought to cause damage in the bowel leading to the symptoms of Crohn's disease.

Patients who complete this study may be eligible for long-term natalizumab therapy via extension protocol ELN100226-351.

ELIGIBILITY:
* Male and female patients at least 18 years of age with at least a six-month history of Crohn's disease and who are currently receiving Remicade and are not in remission (CDAI greater than/equal to 150)
* Women must not be breastfeeding or pregnant, and must not become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-04; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Digestive Disease Associates, Gainesville, Florida
  - Borland Groover Clinic, Jacksonville, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mercury Street Medical, Butte, Montana
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Asheville Gastroenterology, Asheville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - Columbia Gastroenterology Associates, Columbia, South Carolina
  - Gastroenterology Center of the MidSouth, Memphis, Tennessee
  - Memphis Gastroenterology Group, Memphis, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - Internal Medicine Associates, Danville, Virginia
  - Gastroenterology Consultants, Virginia Beach, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Digestive Health Specialists, Tacoma, Washington